CLINICAL TRIAL: NCT03738345
Title: The Effects of Flow Settings During High Flow Nasal Cannula for Adult Hypoxemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HFNC-Flow-003
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hypoxemia
Keywords: High flow nasal cannula; Hypoxemia; Flow setting
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will be masked by the flow setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygenation on hypoxemia patients (Experimental): Adult patients with hypoxemia will be recruited, their own breathing profiles (inspiratory flow, respiratory rates and tidal volume) will be measured. Then patients will be placed on high flow nasal cannula (HFNC), HFNC flow will be titrated based on the hospital's policy or protocol and patient's comfort, patient's clinical effects on oxygenation will be monitored and recorded during the titration process.
  Interventions: Other: HFNC flow
- Lung expansion on healthy volunteer (Experimental): Adult healthy volunteers will be recruited, their own breathing profiles (inspiratory flow, respiratory rates and tidal volume) will be measured. Then they will be placed on HFNC, HFNC flow will be increased sequentially by research protocol and their comfort, subjects' lung expansion effects in different flow will be quantified by Electrical impedance tomography (EIT), a noninvasive assessment tool. Their comfort will also be assessed using a visual scale.
  Interventions: Other: HFNC flow

INTERVENTIONS:
Other: HFNC flow — HFNC flow will be titrated based on the hospital's policy or protocol for hypoxemic patients and research protocol for healthy volunteers

SUMMARY:
High flow nasal cannula (HFNC) delivers oxygen at a flow which exceeds the patient's inspiratory flow demand in order to improve oxygenation. Numerous randomized control trials and meta-analyses have shown that HFNC improves oxygenation and helps avoid intubation in hypoxemic patients, as well as reduce work of breathing, improve ventilation, and decrease hypercapnia in COPD patients. Flow settings play a critical role when using HFNC, as increased flow can reduce inspiratory effort, improve ventilation, and dynamic lung compliance. However, flow rates used in many studies vary widely. The clinical effects of different HFNC flow setting, specifically to match or over than a patients' own inspiratory flow, is still unknown.

DETAILED DESCRIPTION:
High flow nasal cannula (HFNC) delivers oxygen at a flow which exceeds the patient's inspiratory flow demand in order to improve oxygenation. Numerous randomized control trials and meta-analyses have shown that HFNC improves oxygenation and helps avoid intubation in hypoxemic patients, as well as reduce work of breathing, improve ventilation, and decrease hypercapnia in COPD patients. Flow settings play a critical role when using HFNC, as increased flow can reduce inspiratory effort, improve ventilation, and dynamic lung compliance. However, flow rates used in many studies vary widely, from 20-40 LPM in COPD patients and 30-60 LPM in hypoxemic patients. The clinical effects of different HFNC flow setting, specifically to match or over than a patients' own inspiratory flow, is still unknown.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (Age > 18yrs and < 90yrs) who need nasal cannula oxygen flow ≥ 5 L/min to maintain SpO2 at 90-97%.

Exclusion Criteria (Common): - Unable to use resuscitation mask, such as facial trauma, claustrophobia

* Inability to verbally communicate;
* Pregnant
* Inability to breathe via nose, such as nasosinusitis, stuffy nose or nasal obstruction, etc.
* Ordered SpO2 goal is above 97%
* FIO2 needs ≤ 0.4
* Using inhaled pulmonary vasodilator via HFNC

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
SpO2/FIO2 increment for hypoxemic patients | 30 minutes
  SpO2/FIO2 at the optimal/maximum /tolerable/ HFNC flow setting compared to the SpO2/FIO2 at HFNC flow matching patient's inspiratory flow or 30 L/min for hypoxemic patients
RR change for hypoxemic patients | 30 minutes
  Respiratory rates at the optimal/maximum /tolerable/ HFNC flow setting compared to the SpO2/FIO2 at HFNC flow matching patient's inspiratory flow or 30 L/min for hypoxemic patients

SECONDARY OUTCOMES:
comfort scores | 30 minutes
  comfort will be self-evaluation using a visual analog scale with measured score of 0 is the worst and 10 is the best

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after deidentification that underlie the reports reported in this article can be obtained by contacting the corresponding author. Data will be available immediately following publication and ending in 5 years.
Supporting Information: Study Protocol
Time Frame: 5 years following publication
Access Criteria: contacting the corresponding author with clear description on the use of the data

REFERENCES:
- [Result] Ni YN, Luo J, Yu H, Liu D, Ni Z, Cheng J, Liang BM, Liang ZA. Can High-flow Nasal Cannula Reduce the Rate of Endotracheal Intubation in Adult Patients With Acute Respiratory Failure Compared With Conventional Oxygen Therapy and Noninvasive Positive Pressure Ventilation?: A Systematic Review and Meta-analysis. Chest. 2017 Apr;151(4):764-775. doi: 10.1016/j.chest.2017.01.004. Epub 2017 Jan 13. PMID 28089816
- [Result] Pisani L, Fasano L, Corcione N, Comellini V, Musti MA, Brandao M, Bottone D, Calderini E, Navalesi P, Nava S. Change in pulmonary mechanics and the effect on breathing pattern of high flow oxygen therapy in stable hypercapnic COPD. Thorax. 2017 Apr;72(4):373-375. doi: 10.1136/thoraxjnl-2016-209673. Epub 2017 Jan 19. PMID 28104830
- [Result] Mauri T, Alban L, Turrini C, Cambiaghi B, Carlesso E, Taccone P, Bottino N, Lissoni A, Spadaro S, Volta CA, Gattinoni L, Pesenti A, Grasselli G. Optimum support by high-flow nasal cannula in acute hypoxemic respiratory failure: effects of increasing flow rates. Intensive Care Med. 2017 Oct;43(10):1453-1463. doi: 10.1007/s00134-017-4890-1. Epub 2017 Jul 31. PMID 28762180
- [Result] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Result] Delorme M, Bouchard PA, Simon M, Simard S, Lellouche F. Effects of High-Flow Nasal Cannula on the Work of Breathing in Patients Recovering From Acute Respiratory Failure. Crit Care Med. 2017 Dec;45(12):1981-1988. doi: 10.1097/CCM.0000000000002693. PMID 28857852
- [Derived] Li J, Scott JB, Fink JB, Reed B, Roca O, Dhand R. Optimizing high-flow nasal cannula flow settings in adult hypoxemic patients based on peak inspiratory flow during tidal breathing. Ann Intensive Care. 2021 Nov 27;11(1):164. doi: 10.1186/s13613-021-00949-8. PMID 34837553